CLINICAL TRIAL: NCT01853319
Title: An Open-label Phase III Study of Regorafenib in Patients With Metastatic Colorectal Cancer (mCRC) Who Have Progressed After Standard Therapy
Brief Title: Regorafenib in Subjects With Metastatic Colorectal Cancer (mCRC) Who Have Progressed After Standard Therapy
Acronym: REGARD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16754
Record Dates: First submitted 2013-05-06; First posted 2013-05-15 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Neoplasms
Keywords: Regorafenib; Metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regorafenib (Experimental): Regorafenib, 40 mg tablets
  Interventions: Drug: Regorafenib (Stivarga, BAY73- 4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73- 4506) — 160 mg regorafenib per oral every day for 3 weeks of every 4 week cycle (i.e., 3 weeks on, 1 week off)

SUMMARY:
This is an open-label phase III study of regorafenib in patients with metastatic colorectal cancer (mCRC) who have progressed after all approved standard therapy. The purpose of this study is to provide additional information about the safety profile of Regorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects >/= 18 years of age
* Life expectancy of at least 3 months
* Histological or cytological documentation of adenocarcinoma of the colon or rectum
* Subjects with metastatic colorectal cancer (Stage IV)
* Progression during or within 3 months following the last administration of approved standard therapies which must include fluoropyrimidine, oxaliplatin, irinotecan, bevacizumab and cetuximab/panitumumab if KRAS WT (WT: wild-type i.e. no KRAS mutation)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of </= 1
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements
* Women of childbearing potential and men must agree to use adequate contraception since signing of the inform consent (IC) form until at least 3 months after the last study drug administration

Exclusion Criteria:

* Prior treatment with regorafenib
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study drug
* Pregnant or breast-feeding subjects
* Congestive heart failure >/= New York Heart Association (NYHA) class 2
* Myocardial infarction less than 6 months before start of study drug
* Ongoing infection > Grade 2 Common Terminology Criteria for Adverse Events (CTCAE) v. 4.0
* Renal failure requiring hemo-or peritoneal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-07-24 (Actual); Primary Completion 2015-04-24 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 6 months
Number of participants with adverse events which caused withdrawal, dose reduction, interruption or discontinuation | Up to 6 months
Number of death | Up to 6 months
Number of participants with serious adverse events as a measure of safety and tolerability | Up to 6 months
Progression-Free Survival (PFS) | Up to 6 months
  The PFS is defined as the time from date of treatment assignment (i.e., date of first treatment) to date of first observed disease progression or death due to any cause, if death occurs while the subject is in the study (that is, by the last visit including during the safety follow-up visit date), and before progression is observed.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- Turkey (Türkiye) (9):
  - Ankara
  - Antalya
  - Balcali/Adana
  - Bursa
  - Gaziantep
  - Istanbul
  - Izmir
  - Kayseri
  - Samsun

REFERENCES:
- [Derived] Dane F, Ozgurdal K, Yalcin S, Benekli M, Aykan NF, Yucel I, Ozkan M, Evrensel T, Sevinc A, Coskun HS, Sanli UA, Kara IO, Yumuk PF. Safety and efficacy of regorafenib in patients with treatment-refractory metastatic colorectal cancer in Turkey: the single-arm, open-label REGARD study. BMJ Open. 2020 Mar 26;10(3):e027665. doi: 10.1136/bmjopen-2018-027665. PMID 32220908